CLINICAL TRIAL: NCT07146633
Title: Efficacy and Feasibility of Autonomous Eye Movement Desensitization and Reprocessing (A-EMDR) for Patients With Posttraumatic Stress Disorder (PTSD) and Substance Use Disorders
Brief Title: Efficacy of an EMDR App for PTSD and SUD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 167-2023
Record Dates: First submitted 2025-08-13; First posted 2025-08-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Substance Use Disorders
Keywords: EMDR; PTSD; substance dependence
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-EMDR (Experimental)
  Interventions: Behavioral: A-EMDR
- Regular care (Placebo Comparator)
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: A-EMDR — Participants in the treatment group will receive Autonomous Eye movement desensitization and reprocessing (A-EMDR) therapy delivered through an app on their device. Participants will be asked to complete 3 sessions per week for 4 consecutive weeks. During the treatment period, participants will also attend clinical sessions which will focus on factors such as the therapeutic alliance, assessing the participant's current state, reviewing recent alcohol and drug use, reviewing PTSD symptoms, providing a brief counseling intervention, enhancing positive expectancies, inspiring hope, and encouraging adherence to the study protocol.
  Arms: A-EMDR
Other: Treatment as Usual (TAU) — Participants are advised to continue seeking mental health care as usual and will be added to a waitlist for A-EMDR. They will also attend two clinical sessions. Sessions may last 15 to 60 minutes and will focus on factors such as the therapeutic alliance, assessing the participant's current state, reviewing recent alcohol and drug use, reviewing PTSD symptoms, providing a brief counseling intervention, enhancing positive expectancies, inspiring hope, and encouraging adherence to the study protocol. Participants will continue to receive any usual healthcare services as per local standard of care. TAU and other medical appointments will be checked for attendance throughout the study period.
  Arms: Regular care

SUMMARY:
The current proposal is aimed to confirm the efficacy of this novel therapeutic method (autonomous eye movement desensitization and reprocessing; A-EMDR) in a patient group (PTSD and SUD), and to assess the feasibility of the application within this group. While there is no basis to assume lower efficacy of the treatment with this population, confirming that hypothesis is an important and helpful step before a full-performance research study can be initiated. Furthermore, this study proposal will provide additional information regarding the feasibility for this population, which will allow for a more tailored approach in future study.

DETAILED DESCRIPTION:
This is an open-label pilot randomized, wait-list controlled trial evaluating A-EMDR for the treatment of PTSD in patients with SUD for four weeks with a follow up at week eight. Primary outcomes will be measured at the end of the study (week 4) for both groups and at follow up (week 8) for the A-EMDR group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-years old or older
* Fluent in English
* Diagnosed with PTSD by the PTSD Checklist for DSM-5 (PCL-5 past month version score >32)
* Diagnosed with past-year substance use disorder other than caffeine by structured clinical interview for DSM-5 (SCID-5)
* Agrees not to participate in other treatments during the study duration (e.g., mindfulness, yoga, biofeedback, self-hypnosis or tai chi) except individuals who have been already on continuous therapies for at least three months

Exclusion Criteria:

* Diagnosis of a severe or unstable mental illness that precludes safe participation in the study by a healthcare practitioner such as acute psychosis or mania diagnosed by a healthcare practitioner
* Current suicidality risk as indicated during the conduct of the Columbia Suicide Severity Rating Scale (C-SSRS) (21) with concurrence after a study physician's evaluation if the response to C-SSRS questions 1 or 2 is "yes"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in PTSD symptoms and alcohol/drug consumption during 4 weeks of treatment. | From enrollment to the end of treatment at 4 weeks
  We will monitor changes in PTSD symptoms using the clinician-administered PTSD Scale DSM-5 (CAPS-5)/PTSD checklist for DSM-5 (PCL-5) from baseline to weeks four and eight. We will monitor overall alcohol and drug consumption and cravings using the TLFB and CEQ, respectively, over the eight weeks period. In line with previous studies, we will use the Brief Coping Orientation to Problems Experienced (COPE) and subjective measures of substance use coping questionnaire (i.e., How many times have you used a problematic substance for trauma-related problems in the last week? 1) to evaluate the exact frequency of substance used for coping with trauma-related problems from baseline to weeks four and eight. The change in these outcomes will be compared between the A-EMDR and TAU groups.

SECONDARY OUTCOMES:
The feasibility and engagement of A-EMDR during 4 weeks of treatment. | From enrollment to the end of the treatment at 4 weeks
  We will assess the feasibility and engagement of A-EMDR by evaluating the rate of retention (number of participants enrolled after deemed eligible, number of sessions completed for each participant, number of participants who withdraw and/or lost-to-follow-up after enrollment in the study) in the group over the four-week treatment period. We will assess acceptability using quantitative scales to determine their satisfaction with the treatment at weeks four and eight.

CONTACTS AND LOCATIONS:
Locations (1):
- 100 Stokes St, Toronto, Ontario, Canada